CLINICAL TRIAL: NCT00089505
Title: Optimal Combination Therapy After Nevirapine Exposure
Brief Title: NNRTI vs PI Regimens for HIV Infected Women After They Have Taken Nevirapine to Prevent Mother-To-Child HIV Transmission
Acronym: OCTANE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5208; 1U01AI068636 (NIH); OCTANE
Record Dates: First submitted 2004-08-05; First posted 2004-08-06 (Estimated); Results first posted 2011-02-04 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; Treatment Naive; MTCT; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Lopinavir; Nevirapine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- NVP/NVP (Experimental): For participants who had SD NVP exposure prior to study entry. FTC, TDF, and NVP daily the first 14 days, then twice daily. FTC and TDF may be replaced by the combination drug FTC/TDF. Participants who discontinue NVP will receive LPV/RTV twice daily plus two more NRTIs.
  Interventions: Drug: Emtricitabine; Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Nevirapine; Drug: Tenofovir disoproxil fumarate
- NVP/LPV_r (Experimental): For participants who had SD NVP exposure prior to study entry. FTC and TDF daily and LPV/RTV twice daily. FTC and TDF may be replaced by the combination drug FTC/TDF. Participants who discontinue LPV/RTV will receive NVP daily for 14 days before taking it twice daily. plus 2 more NRTIs.
  Interventions: Drug: Emtricitabine; Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Lopinavir/Ritonavir; Drug: Tenofovir disoproxil fumarate
- NoNVP/NVP (Experimental): For participants who did NOT have SD NVP exposure prior to study entry.FTC, TDF, and NVP daily the first 14 days, then twice daily. FTC and TDF may be replaced by the combination drug FTC/TDF. Participants who discontinue NVP will receive LPV/RTV twice daily plus two more NRTIs.
  Interventions: Drug: Emtricitabine; Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Nevirapine; Drug: Tenofovir disoproxil fumarate
- NoNVP/LPV_r (Experimental): For participants who did NOT have SD NVP exposure prior to study entry. FTC and TDF daily and LPV/RTV twice daily. FTC and TDF may be replaced by the combination drug FTC/TDF. Participants who discontinue LPV/RTV will receive NVP daily for 14 days before taking it twice daily. plus 2 more NRTIs.
  Interventions: Drug: Emtricitabine; Drug: Emtricitabine/Tenofovir disoproxil fumarate; Drug: Lopinavir/Ritonavir; Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Emtricitabine — 200 mg taken orally
  Other Names: FTC
Drug: Emtricitabine/Tenofovir disoproxil fumarate — 200/300 mg taken orally
  Other Names: FTC/TDF
Drug: Lopinavir/Ritonavir — 400/100 mg taken orally
  Other Names: LPV/RTV
  Arms: NVP/LPV_r; NoNVP/LPV_r
Drug: Nevirapine — 200 mg taken orally
  Other Names: NVP
  Arms: NVP/NVP; NoNVP/NVP
Drug: Tenofovir disoproxil fumarate — 300 mg taken orally
  Other Names: TDF

SUMMARY:
Non-nucleoside reverse transcriptase inhibitors (NNRTIs) are commonly included in anti-HIV drug regimens. However, HIV infected women who have previously taken the single dose NNRTI nevirapine (SD NVP) for the prevention of mother-to-child transmission (MTCT) of HIV may not respond as well to NNRTIs as women who have never taken NVP. Another class of anti-HIV drugs, protease inhibitors (PIs), may be more effective for women who have previously taken NNRTIs. This study will compare the effectiveness of NNRTI- and PI-based regimens in women who have taken NVP for prevention of MTCT of HIV. This study will also compare regimens including an NNRTI with regimens including a PI in women who have never taken NVP.

DETAILED DESCRIPTION:
NVP is the NNRTI of choice to prevent MTCT of HIV, especially in resource-limited settings. However, prolonged use of NVP may result in drug resistance, decreasing the efficacy of future anti-HIV regimens containing NVP. PIs are more expensive and cause different adverse effects than NNRTIs, but PI-containing regimens may be more effective than NNRTI-containing regimens in treating HIV infected women who previously took NVP for MTCT prophylaxis. This study will compare the efficacy of NNRTI- and PI-containing anti-HIV regimens in women who have previously taken NVP for MTCT of HIV and in women who have never taken NVP.

The study will last a minimum of 48 weeks. Participants will be grouped by previous NVP exposure: participants who have previously taken NVP as MTCT prophylaxis (Trial 1 participants), and participants who have never taken NVP (Trial 2 participants). Participants in each trial will be randomly assigned to one of two arms, NVP-containing arm(NVP/NVP for trial 1 participants and NoNVP/NVP for trial 2 participants) or PI-containing arm(NVP/LPV_r for Trial 1 participants and NoNVP/LPV_r for Trial 2 participants). At the start of the study, Arm NVP/NVP and NoNVP/NVP participants will receive emtricitabine (FTC) daily, tenofovir disoproxil fumarate (TDF) daily, and NVP daily for the first 14 days and then twice daily. Arm NVP/LPV_r and NoNVP/LPV_r participants will receive both FTC and TDF daily and lopinavir/ritonavir (LPV/RTV) twice daily. FTC and TDF may be replaced in either arm with the combination drug FTC/TDF.

If participants experience virologic failure, toxicity, or otherwise cannot tolerate their regimens, they will switch to a different regimen. Arm NVP/NVP and NoNVP/NVP participants will switch to a regimen of two or more nucleoside reverse transcriptase inhibitors (NRTIs) and LPV/RTV; Arm NVP/LPV_r and NoNVP/LPV_r participants will switch to a regimen of two or more NRTIs and NVP. Study visits will occur at entry and at Weeks 2, 4, 8, 12, 16, 24, and then every 12 weeks thereafter. Visits will consist of a physical exam, medication assessment, and blood collection. Participants will be asked to complete adherence questionnaires at Weeks 4, 12, 24, and every 24 weeks thereafter, and quality of life questionnaires at Weeks 24 and ever 24 weeks thereafter. Study drugs will be provided for all participants through 48 weeks after the final participant is randomized.

As per an amendment (dated April 13, 2009), participants will be asked to take part in an extension of this study. Enrollment in the extension is completely voluntary. The purpose of the extension is to monitor, in greater extent, the participants' health as they transition from study treatment to local, clinical care. During the study extension participants will not receive any medications through the study; it is expected that participants will receive their treatments through a local clinic.

Participants enrolling in the extension will enter the extension at the same time as their last visit in the current study. For the extension, participants will be asked to come back to the clinic two times for study visits: at 12 and 72 weeks after entry into the extension. Because there will be a long time between these study visits, participants will also be contacted by phone (or through some other means) close to 48 weeks after entry into the extension.

At each of these visits, participants will be asked about their health and medications, including current anti-HIV drugs. Participants will also be asked about any HIV care received outside of the study. As part of this study, investigators may need to review participants' non-study medical records and speak with their non-study care providers, to find out more about their HIV care and medical problems, and also to check results of lab tests.

During the study extension period, participants will have blood drawn and also be tested for pregnancy.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* HIV infected
* CD4 count less than 200 cells/mm^3 within 90 days prior to study entry
* Plasma HIV-1 RNA using standard Roche Amplicor HIV-1 Monitor Assay within 45 days prior to study entry
* the following laboratory values obtained within 45 days prior to study entry: absolute neutrophil count>=750/mm^3;Hemoglobin>=7.0g/dL;platelet count>=50000/mm^3;aspartate aminotransferase (AST),Alanine aminotransferase (ALT), and alkaline phosphatase <=2.5 x ULN; total bilirubin <=2.5 x ULN
* Normal renal function within 45 days prior to study entry
* Willing to use acceptable forms of contraception
* Karnofsky performance score >=70 on at least one occasion within 45 days prior to study entry
* Parent or guardian willing to provide informed consent, if applicable
* Planning to remain in the same geographical area of residence and are willing to attend study visits as required

Inclusion Criteria for Trial 1 Participants:

* Previously received NVP for prevention of MTCT of HIV
* Has documentation of all prior doses of NVP used for prevention of MTCT of HIV
* Last dose of NVP for prevention of MTCT of HIV taken at least 6 months prior to study entry

Exclusion Criteria for All Participants:

* Previously received any antiretrovirals, excluding NVP for MTCT prophylaxis for Trial 1 participants. Participants who have received up to 10 weeks of zidovudine alone and completed this course at least 6 months prior to study entry are not excluded.
* Use of systemic cancer chemotherapy, systemic investigational agents, immunomodulators, or rifampin within 30 days of study entry
* Pregnant or breastfeeding
* Known allergy or sensitivity to study drugs or their formulations
* Any condition, including drug or alcohol abuse, that, in the opinion of the investigator, may interfere with adherence to study regimens
* Serious illness requiring systemic treatment or hospitalization. Participants who complete therapy or are clinically stable on therapy for at least 30 days prior to study entry are not excluded.
* Tuberculosis (TB) treatment within 30 days prior to study entry
* Use of any prohibited medications within 30 days prior to study entry
* Involuntary incarceration in a correctional facility, prison, or jail for legal reasons or in a medical facility for treatment of either a psychiatric or physical illness

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 745 (Actual)
Dates: Start 2006-11; Primary Completion 2010-08 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahin Lockman, MD, MSc, Study Chair — Brigham and Women's Hospital and Infectious Diseases Division, Department of Immunology and Infectious Diseases, Harvard School of Public Health; Frederick Sawe, MD, Study Chair — The Walter Reed Project/WRAIR
Locations (11):
- Botswana (2):
  - The Gaborone BHP Study Clinic, Bontleng, Gaborone
  - Molepolole BHP Study Clinic, Scottish Livingstone Hospital, Bontleng Gaborone
- Kenya (2):
  - Moi University International Clnical Trials Unit, Eldoret
  - KMRI / Walter Reed Project Clinical Research Center, Kericho
- University of North Carolina Project (UNC Project), Lilongwe, Malawi
- South Africa (3):
  - University of KwaZulu Natal, Durban, KwaZulu-Natal
  - Chris Hani Baragwanath Hospital, Johannesburg, Johannesburg
  - University of Witwatersrand, Johannesburg
- Joint Clinical Research Centre (JCRC), Kampala, Uganda
- Centre for Infectious Disease Research in Zambia (CIDRZ), Lusaka, Zambia
- University of Zimbabwe, Avondale, Harare, Zimbabwe

REFERENCES:
- [Background] Eshleman SH, Jackson JB. Nevirapine resistance after single dose prophylaxis. AIDS Rev. 2002 Apr-Jun;4(2):59-63. PMID 12152519
- [Background] Eshleman SH, Mracna M, Guay LA, Deseyve M, Cunningham S, Mirochnick M, Musoke P, Fleming T, Glenn Fowler M, Mofenson LM, Mmiro F, Jackson JB. Selection and fading of resistance mutations in women and infants receiving nevirapine to prevent HIV-1 vertical transmission (HIVNET 012). AIDS. 2001 Oct 19;15(15):1951-7. doi: 10.1097/00002030-200110190-00006. PMID 11600822
- [Background] Harris M. Efficacy and durability of nevirapine in antiretroviral-experienced patients. J Acquir Immune Defic Syndr. 2003 Sep;34 Suppl 1:S53-8. doi: 10.1097/00126334-200309011-00008. PMID 14562858
- [Background] Jourdain G, Ngo-Giang-Huong N, Le Coeur S, Bowonwatanuwong C, Kantipong P, Leechanachai P, Ariyadej S, Leenasirimakul P, Hammer S, Lallemant M; Perinatal HIV Prevention Trial Group. Intrapartum exposure to nevirapine and subsequent maternal responses to nevirapine-based antiretroviral therapy. N Engl J Med. 2004 Jul 15;351(3):229-40. doi: 10.1056/NEJMoa041305. Epub 2004 Jul 9. PMID 15247339
- [Background] Nightingale S, Dabis F. Evidence behind the WHO guidelines: hospital care for children: what antiretroviral agents and regimens are effective in the prevention of mother-to-child transmission of HIV? J Trop Pediatr. 2006 Aug;52(4):235-8. doi: 10.1093/tropej/fml033. No abstract available. PMID 16877674
- [Background] Turner D, Wainberg MA. HIV transmission and primary drug resistance. AIDS Rev. 2006 Jan-Mar;8(1):17-23. PMID 16736948
- [Derived] Boltz VF, Shao W, Bale MJ, Halvas EK, Luke B, McIntyre JA, Schooley RT, Lockman S, Currier JS, Sawe F, Hogg E, Hughes MD, Kearney MF, Coffin JM, Mellors JW. Linked dual-class HIV resistance mutations are associated with treatment failure. JCI Insight. 2019 Oct 3;4(19):e130118. doi: 10.1172/jci.insight.130118. PMID 31487271
- [Derived] Asmelash A, Zheng Y, Kaloustian KW, Shaffer D, Sawe F, Ogwu A, Salata R, Currier J, Hughes MD, Lockman S. Predictors of suboptimal CD4 response among women achieving virologic suppression in a randomized antiretroviral treatment trial, Africa. BMC Infect Dis. 2014 Jun 17;14:331. doi: 10.1186/1471-2334-14-331. PMID 24938526
- [Derived] Boltz VF, Bao Y, Lockman S, Halvas EK, Kearney MF, McIntyre JA, Schooley RT, Hughes MD, Coffin JM, Mellors JW; OCTANE/A5208 Team. Low-frequency nevirapine (NVP)-resistant HIV-1 variants are not associated with failure of antiretroviral therapy in women without prior exposure to single-dose NVP. J Infect Dis. 2014 Mar 1;209(5):703-10. doi: 10.1093/infdis/jit635. Epub 2014 Jan 16. PMID 24443547
- [Derived] Lockman S, Hughes M, Sawe F, Zheng Y, McIntyre J, Chipato T, Asmelash A, Rassool M, Kimaiyo S, Shaffer D, Hosseinipour M, Mohapi L, Ssali F, Chibowa M, Amod F, Halvas E, Hogg E, Alston-Smith B, Smith L, Schooley R, Mellors J, Currier J; OCTANE (Optimal Combination Therapy After Nevirapine Exposure) ACTG A5208/OCTANE Study Team. Nevirapine- versus lopinavir/ritonavir-based initial therapy for HIV-1 infection among women in Africa: a randomized trial. PLoS Med. 2012;9(6):e1001236. doi: 10.1371/journal.pmed.1001236. Epub 2012 Jun 12. PMID 22719231
- [Derived] Skinner-Adams TS, Butterworth AS, Porter KA, D'Amico R, Sawe F, Shaffer D, Siika A, Hosseinipour MC, Stringer E, Currier JS, Chipato T, Salata R, Lockman S, Eron JJ, Meshnick SR, McCarthy JS. The frequency of malaria is similar among women receiving either lopinavir/ritonavir or nevirapine-based antiretroviral treatment. PLoS One. 2012;7(4):e34399. doi: 10.1371/journal.pone.0034399. Epub 2012 Apr 3. PMID 22509297
- [Derived] Dong BJ, Zheng Y, Hughes MD, Frymoyer A, Verotta D, Lizak P, Sawe F, Currier JS, Lockman S, Aweeka FT; AIDS Clinical Trials Group Study 5208 Team. Nevirapine pharmacokinetics and risk of rash and hepatitis among HIV-infected sub-Saharan African women. AIDS. 2012 Apr 24;26(7):833-41. doi: 10.1097/QAD.0b013e328351a521. PMID 22301417
- [Derived] Porter KA, Cole SR, Eron JJ Jr, Zheng Y, Hughes MD, Lockman S, Poole C, Skinner-Adams TS, Hosseinipour M, Shaffer D, D'Amico R, Sawe FK, Siika A, Stringer E, Currier JS, Chipato T, Salata R, McCarthy JS, Meshnick SR. HIV-1 protease inhibitors and clinical malaria: a secondary analysis of the AIDS Clinical Trials Group A5208 study. Antimicrob Agents Chemother. 2012 Feb;56(2):995-1000. doi: 10.1128/AAC.05322-11. Epub 2011 Nov 28. PMID 22123685
- [Derived] Lockman S, Hughes MD, McIntyre J, Zheng Y, Chipato T, Conradie F, Sawe F, Asmelash A, Hosseinipour MC, Mohapi L, Stringer E, Mngqibisa R, Siika A, Atwine D, Hakim J, Shaffer D, Kanyama C, Wools-Kaloustian K, Salata RA, Hogg E, Alston-Smith B, Walawander A, Purcelle-Smith E, Eshleman S, Rooney J, Rahim S, Mellors JW, Schooley RT, Currier JS; OCTANE A5208 Study Team. Antiretroviral therapies in women after single-dose nevirapine exposure. N Engl J Med. 2010 Oct 14;363(16):1499-509. doi: 10.1056/NEJMoa0906626. PMID 20942666

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited at 10 sites from 7 African countries: 3 from South Africa, 2 from Kenya, and 1 each in Botswana, Malawi, Uganda, Zambia and Zimbabwe, between November 2006 to July 2008. The Botswana site enrolled participants from two locations.
Pre-assignment Details: HIV-infected, treatment-naive women, at least 13 years of age with CD4+ count<200 cells/mm^3. Four participants were randomized but did not start treatment.
Groups:
- NVP/NVP: For participants had single dose Nevirapine (SD NVP) exposure prior to study entry, Emtricitabine capsules(FTC) 200mg (1 capsule orally), Tenofovir disproxil fumerate (TDF) 300mg (1 tablet orally), and NVP 200mg (1 tablet orally) once daily in the morning for the first 14 days, then twice daily after 14 days. FTC and TDF may be replaced by the combination drug FTC/TDF. Participants who discontinue NVP will receive Lopinovir/Ritonovir (LPV/RTV)400/100mg (3 capsules orally) twice daily plus two more Nucleoside reverse transcriptase inhibitors (NRTIs). Following the review on 6 October 2008, the Data Safety Monitoring Board(DSMB) recommended release of the results from this arm.
- NVP/LPV_r: For participants had SD NVP exposure prior to study entry, FTC 200mg (1 capsule orally) and TDF 300mg (1 tablet orally) daily and LPV/RTV 400/100mg (3 capsules orally) twice daily. FTC and TDF may be replaced by the combination drug FTC/TDF. Participants who discontinue LPV/RTV will receive NVP 200mg (1 tablet orally) daily for 14 days before taking it twice daily. plus 2 more NRTIs. Following the review on 6 October 2008, the DSMB recommended release of the results from this arm.
- NoNVP/NVP: For participants had NO SD NVP exposure prior to study entry, FTC 200mg (1 capsule orally), TDF 300mg (1 tablet orally), and NVP 200mg (1 tablet orally) once daily for the first 14 days, then twice daily after 14 days. FTC and TDF may be replaced by the combination drug FTC/TDF. Participants who discontinue NVP will receive LPV/RTV 400/100mg (3 capsules orally) twice daily plus two more NRTIs.
- NoNVP/LPV_r: For participants had SD NVP exposure prior to study entry, FTC 200mg (1 capsule orally) and TDF 300mg (1 tablet orally) once daily and LPV/RTV 400/100mg (3 capsules orally) twice daily. FTC and TDF may be replaced by the combination drug FTC/TDF. Participants who discontinue LPV/RTV will receive NVP daily 200mg (1 tablet orally) for 14 days before taking it twice daily plus 2 more NRTIs.
Period: Overall Study
Arm/Group | NVP/NVP | NVP/LPV_r | NoNVP/NVP | NoNVP/LPV_r
Started | 121 (2 women never started treatment and per protocol, were not followed and not included in analysis.) | 120 | 249 (2 women never started treatment and per protocol, were not followed and not included in analysis.) | 251
Completed | 112 (The results for NVP/NVP were through database cutoff for DSMB review (by 6 October 2008).) | 118 (The results for NVP/LPV_r were through database cutoff for DSMB review (by 6 October 2008).) | 228 | 230
Not Completed | 9 | 2 | 21 | 21
Not completed — Death | 4 | 1 | 5 | 8
Not completed — Withdrawal by Subject | 3 | 0 | 6 | 6
Not completed — Lost to Follow-up | 1 | 1 | 9 | 7
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVP/NVP | NVP/LPV_r | NoNVP/NVP | NoNVP/LPV_r | Total
Number analyzed (Participants) | 121 | 120 | 249 | 251 | 741
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (5) | 31 (5) | 35 (7) | 35 (8) | 33 (7)
Age, Customized [Number; unit: participants]
  Between 13 and 19 years | 0 | 0 | 0 | 2 | 2
  Between 20 and 29 years | 56 | 49 | 63 | 64 | 232
  Between 30 and 39 years | 59 | 62 | 125 | 124 | 370
  Between 40 and 49 years | 5 | 9 | 54 | 49 | 117
  >=50 years | 1 | 0 | 7 | 12 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 120 | 249 | 251 | 741
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 21 | 23 | 45 | 48 | 137
  Zambia | 12 | 12 | 19 | 21 | 64
  Botswana | 13 | 12 | 33 | 30 | 88
  Uganda | 8 | 9 | 22 | 21 | 60
  Malawi | 14 | 10 | 22 | 22 | 68
  South Africa | 35 | 36 | 69 | 67 | 207
  Zimbabwe | 18 | 18 | 39 | 42 | 117
CD4 count Categorical [Number; unit: participants]
  <50 cells/mm^3 | 14 | 11 | 32 | 36 | 93
  Between 50 to 99 cells/mm^3 | 18 | 23 | 63 | 53 | 157
  Between 100 to 149 cells/mm^3 | 35 | 38 | 65 | 78 | 216
  Between 150 to 199 cells/mm^3 | 37 | 32 | 58 | 57 | 184
  Between 200 to 249 cells/mm^3 | 15 | 12 | 18 | 19 | 64
  Between 250 to 299 cells/mm^3 | 1 | 4 | 9 | 4 | 18
  Between 300 to 349 cells/mm^3 | 1 | 0 | 2 | 2 | 5
  >=350 cells/mm^3 | 0 | 0 | 2 | 2 | 4
CD4 count Continuous [Mean (Standard Deviation); unit: cell/mm^3] | 136 (60) | 135 (61) | 126 (68) | 125 (71) | 129 (67)
Baseline HIV-1 RNA Categorial [Number; unit: participants]
  Between 400 and 999 copies/mL | 0 | 1 | 1 | 2 | 4
  Between 1000 and 9,999 copies/mL | 5 | 8 | 18 | 11 | 42
  Between 10,000 and 99,999 copies/mL | 44 | 33 | 81 | 88 | 246
  Between 100,000 and 749,999 copies/mL | 61 | 63 | 123 | 128 | 375
  >=750,000 copies/mL | 11 | 15 | 26 | 22 | 74
HIV-1 RNA Continuous [Median (Inter-Quartile Range); unit: log 10 copies/mL] | 5.2 [4.3 to 5.8] | 5.1 [4.2 to 5.9] | 5.2 [4.2 to 5.9] | 5.2 [4.3 to 5.8] | 5.2 [4.7 to 5.5]
WHO stage [Number; unit: participants] — World Health Organization (WHO) produced WHO Disease Staging System for HIV Infection and Disease in Adults and Adolescents. It is an approach for use in resource limited settings in studies of progression to symptomatic HIV disease. There are 4 stages of disease staging, 1 being the least severe and 4 being the most severe disease stage based on the HIV related symptoms and diagnoses. Please refer to the following web page for detailed staging criteria: http://www.who.int/docstore/hiv/scaling/anex1.html
  participants
    Clinical stage I | 44 | 56 | 97 | 93 | 290
    Clinical stage II | 42 | 38 | 72 | 67 | 219
    Clinical stage III | 30 | 25 | 73 | 80 | 208
    Clinical stage IV | 5 | 1 | 7 | 11 | 24

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Who Experienced Virologic Failure or Died.
Description: Virologic failure (VF) is defined as a plasma HIV-1 RNA level that is 1 log10 below baseline 12 weeks after treatment is initiated or as a plasma HIV-1 RNA level that is >=400 copies/mL at or after 24 weeks of treatment, regardless of whether randomized treatment was being taken at the time of VF.
Time Frame: Through database cutoff for DSMB review (by October 6, 2008) for NVP/NVP and NVP/LPV_r. Throughout study for NoNVP/NVP and NoNVP/LPV_r.
Population: Numbers presented use the intent-to-treat approach (i.e. ignoring changes from randomized treatment).
Measure: Number; unit: participants
Arm/Group | NVP/NVP | NVP/LPV_r | NoNVP/NVP | NoNVP/LPV_r
Number analyzed (Participants) | 121 | 120 | 249 | 251
participants | 32 | 10 | 42 | 50

2. Secondary Outcome: Percent of Participants Who Experienced Virologic Failure or Died
Description: Results report cumulative percent of participants reaching virologic failure (VF) or death by week 48 and week 96 calculated using the Kaplan-Meier method. VF is defined as a plasma HIV-1 RNA level that is 1 log10 below baseline 12 weeks after treatment is initiated or as a plasma HIV-1 RNA level that is >=400 copies/mL at or after 24 weeks of treatment, regardless of whether randomized treatment was being taken at the time of VF.
Time Frame: Through database cutoff for DSMB review (by October 6, 2008) for NVP/NVP and NVP/LPV_r arms. Throughout study for NoNVP/NVP and NoNVP/LPV_r arms.
Population: Numbers presented use the intent-to-treat approach (i.e. ignoring changes from randomized treatment).
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | NVP/NVP | NVP/LPV_r | NoNVP/NVP | NoNVP/LPV_r
Number analyzed (Participants) | 121 | 120 | 249 | 251
Percent of participants
  week 48 percent of virologic failure or death | 23 [16 to 31] | 4 [1 to 8] | 14 [10 to 19] | 14 [9 to 18]
  week 96 percent of virologic failure or death | 31 [21 to 40] | 12 [5 to 20] | 17 [12 to 21] | 20 [14 to 25]

3. Secondary Outcome: CD4 Count Change From Randomization
Description: Change was calculated as the CD4 count at Week 48 (or at Week 96) minus the baseline CD4 count (last CD4 before/on treatment start date). For NVP/NVP and NVP/LPV_r arms, data through DSMB review cutoff (October 6, 2008) were used to report the outcome. For NoNVP/NVP and NoNVP/LPV_r arms, since the follow-up continued as planned, data through overall study were used.
Time Frame: Through database cutoff for DSMB review (by October 6, 2008) for NVP/NVP and NVP/LPV_r. Throughout study for NoNVP/NVP and NoNVP/LPV_r. Week 48 and 96.
Population: Changes were calculated using the intent-to-treat approach (i.e. ignoring changes from randomized treatment) but no imputation was done for missing values.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | NVP/NVP | NVP/LPV_r | NoNVP/NVP | NoNVP/LPV_r
Number analyzed (Participants) | 121 | 120 | 249 | 251
cells/mm^3
  Week 48 CD4 count change from randomization | 191 [120 to 270] | 201 [142 to 280] | 172 [97 to 246] | 172 [97 to 268]
  Week 96 CD4 count change from randomization | 291 [189 to 366] | 278 [180 to 360] | 223 [142 to 339] | 256 [149 to 379]

4. Secondary Outcome: Number of Participants Who Experienced Treatment-related Toxicity That Led to Discontinuation of Randomized Regimen.
Description: The outcome is defined as treatment-related toxicity (as evaluated by sites), regardless of grade, that led to discontinuation of randomized regimen. For NVP/NVP and NVP/LPV_r arms, data through DSMB review cutoff (October 6, 2008) were used to report the outcome. For NoNVP/NVP and NoNVP/LPV_r arms, since the follow-up continued as planned, data through overall study were used.
Time Frame: as for outcome 1
Population: Numbers presented use as-treated method.
Measure: Number; unit: participants
Arm/Group | NVP/NVP | NVP/LPV_r | NoNVP/NVP | NoNVP/LPV_r
Number analyzed (Participants) | 121 | 120 | 249 | 251
participants | 15 [0.06 to 0.17] | 0 [NA to NA] | 35 [0.09 to 0.18] | 0 [NA to NA]

5. Secondary Outcome: Number of Participants Who Experienced HIV-related Disease Progression or Death
Description: Worsening to WHO stage III/IV (among subjects who had WHO stage I/II at baseline) and death were the composite secondary endpoint. WHO Disease Staging System for HIV Infection and Disease in Adults and Adolescents is an approach for use in resource limited settings in studies of progression to symptomatic HIV disease. There are 4 stages of disease staging, 1 being the least severe and 4 being the most severe disease stage based on the HIV related symptoms and diagnoses. Please refer to the following web page for detailed staging criteria: http://www.who.int/docstore/hiv/scaling/anex1.html
Time Frame: as for outcome 1
Population: Numbers presented use the intent-to-treat approach (i.e. ignoring changes from randomized treatment).
Measure: Number; unit: participants
Arm/Group | NVP/NVP | NVP/LPV_r | NoNVP/NVP | NoNVP/LPV_r
Number analyzed (Participants) | 121 | 120 | 249 | 251
participants | 6 [0.01 to 0.09] | 4 [0.01 to 0.07] | 19 [0.04 to 0.11] | 26 [0.05 to 0.11]

6. Primary Outcome: Time From Randomization to Virologic Failure or Death for Participants Who Had SD NVP Exposure Prior to Study Entry
Description: 5th and 10th Percentiles in weeks from randomization to virologic failure (VF) or death. VF is defined as a plasma HIV-1 RNA level that is 1 log10 below baseline 12 weeks after treatment is initiated or as a plasma HIV-1 RNA level that is >=400 copies/mL at or after 24 weeks of treatment, regardless of whether randomized treatment was being taken at the time of VF.
Time Frame: Through database cutoff for DSMB review (by October 6, 2008) with median follow-up 72 weeks and range from 0 to 144 weeks.
Population: Numbers presented use the intent-to-treat approach (i.e. ignoring changes from randomized treatment).
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | NVP/NVP | NVP/LPV_r | NoNVP/NVP | NoNVP/LPV_r
Number analyzed (Participants) | 121 | 120 | 0 | 0
weeks
  5th percentile | 12 [6 to 12] | 60 [12 to 84] |  |
  10th percentile | 12 [12 to 24] | 84 [60 to NA] — Not estimable as the upper limit for survival function at all weeks is above 90% |  |
  25th percentile | 60 [24 to NA] — Not estimable as the upper limit for survival function at all weeks is above 75% | NA [NA to NA] — Not estimable as the estimates for survival function at all weeks is above 75% |  |
Statistical Analysis 1: Comparison: NVP/NVP vs NVP/LPV_r; Test type: Superiority or Other; p < 0.001, Regression, Cox — P-value was not adjusted for multiple interim analyses, but any adjustment would be negligible because Peto-Haybittle spending function was used as a basis for calculating the repeated confidence intervals used in interim monitoring; The model was stratified by screening CD4 strata (<50 vs. >=50 cells/mm^3); Hazard Ratio (HR) = 3.69, 95% CI 2-sided [1.79 to 7.61] — The HR is for NVP/NVP vs. NVP/LPV_r

7. Primary Outcome: Time From Randomization to Virologic Failure or Death for Participants Without SD NVP Exposure Prior to Study Entry
Description: as for outcome 6
Time Frame: Throughout study with median follow-up 72 weeks and range from 0 to 180 weeks.
Population: The analysis was intent to treat per protocol.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | NVP/NVP | NVP/LPV_r | NoNVP/NVP | NoNVP/LPV_r
Number analyzed (Participants) | 0 | 0 | 249 | 251
weeks
  5th percentile |  |  | 24 [12 to 24] | 12 [12 to 24]
  10th percentile |  |  | 36 [24 to 48] | 36 [12 to 60]
  25th percentile |  |  | NA [120 to NA] — Not estimable as the estimate for survival function at all weeks is above 75% | 132 [96 to NA] — Not estimable as the upper limit for survival function at all weeks is above 75%
Statistical Analysis 1: Comparison: NoNVP/NVP vs NoNVP/LPV_r; Test type: Non-Inferiority or Equivalence — NoNVP/NVP regimen will be considered equivalent to the NoNVP/LPV_r regimen if the two-sided 95% confidence interval for the hazard ratio for virologi falure is entirely below 2.0; equivalence will be established if the same confidence interval is entirely within the range 0.5 to 2.0; p = 0.43, Regression, Cox — P-value is for a test of superiority and was not adjusted for interim analyses, but any adjustment would be negligible because Peto-Haybittle spending function was used as a basis for calculating the repeated confidence intervals used; The cox proportional hazard model was stratified by screening CD4 strata (<50 vs. >=50 cells/mm3); Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.56 to 1.29] — The HR is for NoNVP/NVP vs. NoNVP/LPV_r

8. Secondary Outcome: Number of Participants Who Received NVP-containing Regimens at Randomization and Experienced NVP-associated Rash or Grade 2+ Liver Lab Abnormality
Description: Any grade of rash or grade 2+ liver lab abnormality events that were claimed to be NVP associated (definitely, probably, or possibly) by site investigators were evaluated. Grade 2+ liver lab abnormality is defined as aspartate aminotransferase (AST)>=2.6 x ULN or alanine aminotransferase (ALT)>=2.6 x ULN.
Time Frame: Through database cutoff for DSMB review (by October 6, 2008) for NVP/NVP arm. Throughout study for NoNVP/NVP arm.
Population: Numbers presented use the as-treated approach.
Measure: Number; unit: participants
Arm/Group | NVP/NVP | NVP/LPV_r | NoNVP/NVP | NoNVP/LPV_r
Number analyzed (Participants) | 121 | 0 | 249 | 0
participants | 20 |  | 51 |

9. Secondary Outcome: Percent of Participants Who Reported to Never Missed Any of the Study Drug Regimen in the Past Month
Description: Self-reported adherence at week 48 and 96 while participants remained on randomized regimen. Adherence interviews for each antiretroviral drug drug the participant is taking was performed by site personnel every 24 weeks. For NVP/NVP and NVP/LPV_r arms, data through DSMB review cutoff (October 6, 2008) were used to report the outcome. For NoNVP/NVP and NoNVP/LPV_r arms, since the follow-up continued as planned, data through overall study were used.
Time Frame: as for outcome 2
Population: Numbers presented use as-treated approach.
Measure: Number; unit: percent of participants
Arm/Group | NVP/NVP | NVP/LPV_r | NoNVP/NVP | NoNVP/LPV_r
Number analyzed (Participants) | 121 | 120 | 249 | 251
percent of participants
  week 48 percent of full adherence in past month | 89 | 88 | 90 | 86
  week 96 percent of full adherence in past month | 94 | 95 | 93 | 87

ADVERSE EVENTS:
Time Frame: Through database cutoff for DSMB review (by October 6, 2008) for NVP/NVP and NVP/LPV_r arms (with median follow-up: 72 weeks; range 0 -144 weeks). Throughout study for NoNVP/NVP and NoNVP/LPV_r arms (median follow-up: 72 weeks; range 0-180 weeks).
Arm/Group | NVP/NVP | NVP/LPV_r | NoNVP/NVP | NoNVP/LPV_r
Serious Adverse Events (participants affected / at risk) | 9/121 | 6/120 | 26/249 | 19/251
Other Adverse Events (participants affected / at risk) | 110/121 | 105/120 | 225/249 | 227/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVP/NVP (N=121) | NVP/LPV_r (N=120) | NoNVP/NVP (N=249) | NoNVP/LPV_r (N=251)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2
Fanconi syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Abdominal pain uppr (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1 | 2
Death neonatal (General disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 5 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 2
HIV infection (Infections and infestations) | 1 | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 0 | 1 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis tuberculous (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 5 | 3
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Steve-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NVP/NVP (N=121) | NVP/LPV_r (N=120) | NoNVP/NVP (N=249) | NoNVP/LPV_r (N=251)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 | 9 | 17 | 12
Abdominal pain (Gastrointestinal disorders) | 14 | 12 | 22 | 26
Abdominal pain lower (Gastrointestinal disorders) | 3 | 8 | 14 | 18
Diarrhoea (Gastrointestinal disorders) | 15 | 17 | 29 | 38
Nausea (Gastrointestinal disorders) | 10 | 3 | 19 | 23
Vomiting (Gastrointestinal disorders) | 17 | 14 | 33 | 32
Asthenia (General disorders) | 6 | 2 | 7 | 14
Chest pain (General disorders) | 9 | 5 | 30 | 25
Chills (General disorders) | 12 | 12 | 14 | 20
Malaise (General disorders) | 6 | 6 | 10 | 9
Pain (General disorders) | 7 | 8 | 14 | 11 (251)
Pyrexia (General disorders) | 22 | 17 | 52 | 46
Body tinea (Infections and infestations) | 7 | 3 | 10 | 9
Gastroenteritis (Infections and infestations) | 7 | 4 | 13 | 15
Genital herpes (Infections and infestations) | 7 | 5 | 8 | 6
Herpes zoster (Infections and infestations) | 3 | 2 | 13 | 8
Malaria (Infections and infestations) | 21 | 25 | 43 | 43
Oral candidiasis (Infections and infestations) | 6 | 3 | 13 | 15 (251)
Pelvic inflammatory disease (Infections and infestations) | 4 | 6 | 12 | 15
Pneumonia bacterial (Infections and infestations) | 9 | 4 | 21 | 22
Pulmonary tuberculosis (Infections and infestations) | 5 | 5 | 9 | 15
Upper respiratory tract infection (Infections and infestations) | 18 | 15 | 33 | 31
Urinary tract infection (Infections and infestations) | 5 | 6 | 13 | 16
Vulvovaginal cadidiasis (Infections and infestations) | 13 | 15 | 26 | 32
Alanine aminotransferase increased (Investigations) | 23 | 10 | 40 | 20
Aspartate aminotransferase increased (Investigations) | 23 | 12 | 49 | 31
Blookd albumin abnormal (Investigations) | 17 | 15 | 38 | 36
Blood alkaline phosphatase increased (Investigations) | 8 | 1 | 20 | 2
Blood bicarbonate abnormal (Investigations) | 12 | 8 | 26 | 25
Blood cholesterol abnormal (Investigations) | 1 | 3 | 14 | 14
Blood glucose decreased (Investigations) | 7 | 4 | 10 | 4
Blood potassium decreased (Investigations) | 17 | 8 | 6 | 21
Blood sodium decreased (Investigations) | 21 | 24 | 49 | 58
Haemoglobin decreased (Investigations) | 14 | 12 | 38 | 40
Low density lipoprotein (Investigations) | 3 | 5 | 14 | 9
Neutrophil count decreased (Investigations) | 28 | 35 | 68 | 64
Weight decreased (Investigations) | 7 | 10 | 10 | 25
White blood cell count decreased (Investigations) | 11 | 14 | 21 | 33
Decreased appetite (Metabolism and nutrition disorders) | 4 | 6 | 13 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 10 | 15 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | 11 (249) | 14
Headache (Nervous system disorders) | 25 | 31 | 53 | 51
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 6 | 19 | 24
Dysuria (Renal and urinary disorders) | 6 | 7 | 12 | 11
Vaginal discharge (Reproductive system and breast disorders) | 17 | 14 | 45 | 42
Vulvovaginal pruritus (Reproductive system and breast disorders) | 10 | 11 | 19 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 26 | 60 | 55
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 10 | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 15 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 14 | 31 | 34
Rash (Skin and subcutaneous tissue disorders) | 28 | 27 | 66 | 67
Rash papular (Skin and subcutaneous tissue disorders) | 7 | 6 | 20 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.